CLINICAL TRIAL: NCT01083004
Title: A Randomized Study Comparing Brilliant Blue and Indocyanine Green as Intravitreal Dye in Macular Pucker and Macular Hole
Brief Title: Brilliant Blue Versus Indocyanine Green
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Prof. Dr. B. Kirchhof, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BlueIce001
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2007-10

CONDITIONS: Macular Pucker; Macular Hole; Vitreoretinal Surgery
Keywords: dye; internal limiting membrane; macular hole; macular pucker
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations | interventions — Indocyanine Green

ARMS (2):
- Indocyanine green arm (Active Comparator)
  Interventions: Procedure: Indocyanine green
- Brilliant blue (Active Comparator)
  Interventions: Procedure: Brilliant blue arm

INTERVENTIONS:
Procedure: Indocyanine green — Using indocyanine green as intraoperative dye
  Arms: Indocyanine green arm
Procedure: Brilliant blue arm — Using brilliant blue as intraoperative dye
  Arms: Brilliant blue

SUMMARY:
A study of non-inferiority design comparing brilliant blue and indocyanine green as intraoperative dye in macular pucker and macular hole.

ELIGIBILITY:
Inclusion Criteria:

* age over 50
* macular pucker or macular hole with subjective disturbances
* All phakic or pseudophakic patients
* far visual acuity better than 20/400
* able to read, understand, and willing to sign the informed consent form

Exclusion Criteria:

* any other ocular disease or conditions compromising the visual acuity other than macular hole or macular pucker
* prior vitreoretinal surgery in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Best corrected far visual acuity (ETDRS) | 1 year postoperative

SECONDARY OUTCOMES:
Reading ability (Radner) | 1 Year
Optical coherence tomography | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Kirchhof, MD, Principal Investigator — University of Cologne, Center of Ophthalmology, 50924 Cologne, Germany
Locations (1):
- Center of Ophthalmology, University of Cologne, Cologne, North Rhine-Westphalia, Germany